CLINICAL TRIAL: NCT07289854
Title: Portable Endoscopic Camera System Using Modified Action Camera for Endoscopic Sinunasal Examination
Status: Recruiting | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 299385
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Nasolacrimal Duct Obstruction; Nasolacrimal Tract Obstruction
MeSH Terms: conditions — Lacrimal Duct Obstruction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Modified Portable Endoscopic Camera
  Interventions: Device: Modified Portable Endoscopic Camera

INTERVENTIONS:
Device: Modified Portable Endoscopic Camera — The Sony Action Camera was modified to allow direct coupling with a standard rigid nasal endoscope:
  1. The native 180° wide-angle lens was replaced with a narrow-field 31° lens, enabling full-frame capture of the endoscopic image without peripheral distortion.
  2. The camera housing was adapted by attaching a ¾-inch water pipe end connector, serving as a secure and stable mount for the endoscope eyepiece.
  The modified system captures both video and still images.

SUMMARY:
This study is designed to compare two methods for performing a nasal endoscopic examination used in the evaluation of excessive watering or tearing of the eyes. The purpose of the study is to determine whether a new, smaller, modified camera system can produce images of the inside of the nose that are as clear and useful as those produced by the standard endoscopic camera system currently used in clinics.

The study seeks to answer the question of whether a compact, easy-to-store camera system can provide similar diagnostic image quality to the traditional, larger tower-based system. The clinical steps of the nasal examination remain the same; the only difference is the type of camera system used to capture the images.

DETAILED DESCRIPTION:
This study evaluates two imaging systems used during routine nasal endoscopy performed for assessment of epiphora and related nasolacrimal or sinonasal concerns. The protocol involves conducting a standard nasal endoscopic examination with the conventional full-size tower-mounted camera system typically utilized in ophthalmology and otolaryngology outpatient settings, followed by a second examination using a modified compact camera system. Both examinations use the same endoscope and follow identical clinical steps.

The modified camera system attaches at the usual hand-position point on the endoscope and is designed to reduce equipment footprint, increase portability, and simplify storage. The second examination adds an estimated 3-5 minutes to the clinical encounter and does not introduce additional maneuvers or diagnostic procedures.

The primary objective is to compare image quality between the standard system and the compact system. Secondary objectives include assessments of device usability, handling characteristics, and overall feasibility of integrating the compact system into routine clinical workflow.

This evaluation aims to determine whether the compact camera system can provide imaging performance comparable to the traditional tower-based system while offering potential operational benefits. These benefits may include improved flexibility in space-constrained environments, reduced dependence on fixed equipment, and expanded opportunities for nasal endoscopy in clinics with limited infrastructure. Findings may inform future decisions regarding endoscopic equipment selection across various clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older) presenting with tearing suggestive of nasolacrimal drainage obstruction
* Adult patients presenting with sinunasal disease with clinical findings on endonasal examination.
* Adult patients who require a clinically ordered nasal endoscopic exam.

Exclusion Criteria:

* Children (Under the age of 18)
* Patients with over secretory tearing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults receiving care in the ophthalmology or otolaryngology outpatient clinics at the University of Arkansas for Medical Sciences (UAMS) who present with sinonasal or lacrimal tearing symptoms and require nasal endoscopic evaluation as part of routine clinical care. Potential participants will be identified only during their scheduled clinic visits, and no individuals will be contacted in advance. Eligibility confirmation will be based solely on information already available in the medical record during standard outpatient workflow. Individuals who meet eligibility will be approached in person during the clinic visit and invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Image Quality Score of Modified Portable Endoscopic Camera System | Grading completed within 3 months of enrollment completion.
  Image quality of the modified portable endoscopic camera system will be evaluated using a 5-point Likert scale assessing resolution, clarity of anatomical structures, and overall clinical utility. Three attending physicians will independently grade anonymized images from each nasal anatomical site. Scores will be compared with those obtained from the standard endoscopic tower.

SECONDARY OUTCOMES:
Image Quality Score of Standard Endoscopic Tower System | Grading completed within 3 months of enrollment completion.
  Image quality of the standard endoscopic tower will be evaluated using the same 5-point Likert grading scale and process applied to the modified system. These scores will serve as the comparator for paired analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Solyman, MD, Principal Investigator — University Of Arkansas For Medical Sciences, Jones Eye Institute
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT07289854/Prot_SAP_000.pdf